CLINICAL TRIAL: NCT06220994
Title: The Gut Microbiome and Metabolomics Among Chronic Lower Extremities Threatening Ischemia Patients in China - a Prospective Observational Study
Brief Title: the Gut Microbiome and Metabolomics in Chronic Lower extreMities Threatening Ischemia
Acronym: MMM
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 21431-4-01
Record Dates: First submitted 2023-02-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-03

CONDITIONS: Chronic Limb-threatening Ischemia; Microtia
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Congenital Microtia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Peripheral blood plasma and stool.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic limb-threatening ischemia: Resting pain for at least 2 weeks with at least one hemodynamic index: ABI<0.4,AP<50mmHg, TP or TCPO2<30mmHg. Tissue defects (ulceration or gangrene) persisted for at least 2 weeks with at least one significant PAD objective evidence: ABI<0.8, AP<100mmHg, TP or TCPO2<60mmHg.
- health control: sex - and age-matched healthy people (without history of atherosclerotic plaque, coronary heart disease or stroke).

SUMMARY:
Intestinal floras and their metabolites are involved in progressing metabolic and cardiovascular diseases. However, currently, articles related to the relationship between intestinal floras and atherosclerosis mainly focus on coronary atherosclerotic disease (CAD) population, or atherosclerosis model animals such as ApoE-/-, LDLR-/- high-fat diet mice, and there are few studies on Chronic limb-threatening ischemia (CLTI). CLTI and CAD have a similar pathological basis of atherosclerosis. It is unclear whether intestinal flora plays an essential role in the occurrence and development of CLTI. This project aims to explore the relation between microorganisms, metabolites, and CLTI.

DETAILED DESCRIPTION:
This project aims to study the intestinal flora and its metabolites in patients with CLTI, explore whether CLTI patients and CAD patients have their own characteristic flora, analyze the microorganisms and metabolites markers of poor prognosis in patients with CLTI, and screen out the key differential bacteria and metabolites that inhibit the progress of CLTI, in order to provide new insights and research basis for the treatment of CLTI.

ELIGIBILITY:
Inclusion Criteria:

Control group: sex - and age-matched healthy people (without history of atherosclerotic plaque, coronary heart disease or stroke).

Case group: resting pain for at least 2 weeks with at least one hemodynamic index: ABI<0.4,AP<50mmHg, TP or TCPO2<30mmHg. Tissue defects (ulceration or gangrene) persisted for at least 2 weeks with at least one significant PAD objective evidence: ABI<0.8, AP<100mmHg, TP or TCPO2<60mmHg.

Exclusion Criteria:

1. Patients with inflammatory bowel disease, autoimmune diseases, malignancies, infectious diseases, and severe liver and kidney dysfunction (cirrhosis, CKD stage 4 and 5).
2. Patients with thromboembolic angiitis, arterial embolism, and takayasu.
3. Patients who have used probiotics or antibiotics in the last 2 months.
4. After interventional surgery and amputation below the knee or above knee.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Chronic limb-threatening ischemia patients and health adult without history of atherosclerotic plaque, coronary heart disease or stroke, attending Tsinghua Chang Gung Hospital in Beijing.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-11-15 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Bacteria or metabolites associated with prolonged survival time without above-knee amputation | 3years.
  The relationship between the prognosis and gut microbiota or plasma metabolomics was analyzed. Spearman correlations between CAGs, serum metabolite modules and clinical parameters were calculated using R, and both differential abundances of CAGs and CLTI-associated metabotypes were tested by the Wilcoxon rank sum test.

SECONDARY OUTCOMES:
Key bacteria in CLTI | up to 1 week
  Differential bacteria enriched in healthy group but absent in CLTI patients were explored by metagenomic analysis of the gut microbiota. It includes species composition and abundance analysis, beta diversity, differences between groups, and RDA/CCA.
Key plasma metabolites in CLTI | up to 1 week
  Differential metabolites enriched in healthy group but absent in CLTI patients were explored by non-targeted metabolomics analysis of the gut contents. It includes sample grouping data analysis, metabolites annotation, and screening of differential metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Weiwei Wu, MD, Principal Investigator — Beijing Tsinghua Chang Gung Hospital
Locations (1):
- Beijing Tsinghua Chang Gung Hosipital, Beijing, Beijing Municipality, China